CLINICAL TRIAL: NCT01896440
Title: The Effects of Ondansetron on Myocardial Repolarization in Children Receiving Chemotherapy
Brief Title: Heart Safety Study of Ondansetron in Children Receiving Chemotherapy
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: FDA did not approve
Sponsor: University of Oklahoma (Other)
Responsible Party: Principal Investigator, Rene Y McNall-Knapp, MD, Associate Professor, University of Oklahoma
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pediatric ondansetron QTc
Record Dates: First submitted 2013-07-01; First posted 2013-07-11 (Estimated); Last update posted 2013-10-08 (Estimated); Status verified 2013-10

CONDITIONS: Malignant Childhood Neoplasm
Keywords: Pediatric; Ondansetron; Cardiac repolarization; QTc interval
MeSH Terms: conditions — Neoplasms | interventions — Ondansetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A - standard ondansetron dose first (Active Comparator): Group A will receive the standard dose of ondansetron (0.15 mg/kg) with the first cycle of chemotherapy and the high dose (0.3 mg/kg) with second cycle.
  Interventions: Drug: Ondansetron
- Group B - high dose ondansetron first (Active Comparator): Group B patients will receive the higher dose of ondansetron (0.3 mg/kg) with the first cycle of chemotherapy and the standard dose (0.15 mg/kg) with the second.
  Interventions: Drug: Ondansetron

INTERVENTIONS:
Drug: Ondansetron — There will be two doses investigated in each arm - standard dose (0.15 mg/kg) and high dose (0.3 mg/kg)
  Other Names: Zofran

SUMMARY:
We will study the effects of ondansetron on measurements of electrical activity in the heart to make sure doses we are using to prevent nausea and vomiting in children receiving chemotherapy are safe.

DETAILED DESCRIPTION:
Children receiving chemotherapy for cancer at the Jimmy Everest Center for Cancer and Blood Disorders in Children also often receive an IV dose of an antiemetic for prophylaxis. The most common antiemetics used are in the family of 5HT3 antagonists, specifically granisetron and ondansetron. Prior to a recent recommendation by the FDA, we have used ondansetron 0.45 mg/kg IV. Based on adult ECG data, the recommended dose of ondansetron has been changed to no greater than 0.15 mg/kg. We have prior studies showing that the bigger dose is better at preventing nausea and vomiting. Therefore we are studying ECG data in patients receiving ondansetron and chemotherapy. Each subject will have two identical cycles of chemotherapy. Prior to the first of the two cycles they will be randomized to receive one of two doses of ondansetron with the first cycle and the other dose with the second cycle. The two doses are the recommended dose of 0.15 mg/kg and a higher dose of 0.3 mg/kg. The dose level the patient receives each cycle will be blinded to the investigator and the subject.

Prior to the first dose of investigational ondansetron, the patient will have an ECG. This ECG will be repeated 30 minutes after the ondansetron is administered and just before chemotherapy administration, and repeated again 30 minutes later. The change in the QTc intervals will be calculated by two independent pediatric cardiologists who are also blinded to the ondansetron dose level received. This process will be repeated with the next course of chemotherapy, with the second dose of ondansetron. Our goal is to see if there is an appreciable difference between the two doses in the QTc interval changes they induce.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 months to 18 years
* Diagnosis of cancer and receiving 2 identical cycles of chemotherapy within 2 months of each other

Exclusion Criteria:

* History of cardiac conduction anomalies, myocardial infarction, structural heart abnormalities (even if repaired)
* Pregnant or of child-bearing age and unwilling to take a pregnancy test
* Potassium or calcium outside of reference range at screening
* Liver enzymes (AST/ALT) or bilirubin >/= 2 x the upper limit of normal at screening

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2013-10; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Change in QTc interval | Day 1 to 2 months
  QTc intervals will be estimated by performing ECGs on patients pre-investigational drug administration and post-investigational drug administration. The change in the QTc interval between the two ECGs for each investigational dose is the primary endpoint.

CONTACTS AND LOCATIONS:
Overall Officials: Rene Y McNall-Knapp, MD, Principal Investigator — University of Oklahoma; Matthew Campbell, MD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States